CLINICAL TRIAL: NCT03653910
Title: Effect-site Concentration of Remifentanil for Inhibiting Cardiovascular Responses to Double-lumen Tube Intubation With Airtraq Videolaryngoscopy: a Comparative Study With Macintosh Laryngoscopy
Brief Title: Effect-site Concentration of Remifentanil for Double-lumen Tubes Intubation: Airtraq VS Macintosh Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wenlong Yao, M.D,PhD, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJMZK20180713
Record Dates: First submitted 2018-08-06; First posted 2018-08-31 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Hemodynamic Instability; Intubation Complication
Keywords: double-lumen tube intubation; remifentanil; target controlled infusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Airtraq (Experimental): Patients received DLT intubation by Airtraq videolarygoscope
  Interventions: Device: Airtraq
- Macintosh (Active Comparator): Patients received DLT intubation by Macintosh laryngoscope
  Interventions: Device: Macintosh

INTERVENTIONS:
Device: Airtraq — Airtraq is a kind of videolaryngoscope for intubation
  Arms: Airtraq
Device: Macintosh — Macintosh is a traditional laryngoscope for intubation
  Arms: Macintosh

SUMMARY:
The 50% effective concentration of remifentanil by target controlled infusion was not determined for inhibiting the haemodynamic response during double-lumen tube (DLT) intubation. Previous study showed that Airtraq videolaryngoscope provided more stable haemodynamics than Macintosh for double-lumen tube intubation. In this study, the investigators will compare the 50% effective concentration of remifentanil between Airtraq videolaryngoscope and Macintosh laryngoscope for inhibiting haemodynamic responses during DLT intubation.

DETAILED DESCRIPTION:
Dixon "up-and-down" method was used to determine 50% effective concentration of remifentanil by target controlled infusion for inhibiting the haemodynamic responses during DLT intubation with Airtraq videolaryngoscope or Macintosh laryngoscope.

ELIGIBILITY:
Inclusion Criterias:

1. American Society of Anesthesiologists physical status of I-II
2. Patients aged 18-65 years
3. BMI 18-35 kg/m2
4. Elective pulmonary surgery under general anesthesia to double-lumen tubes intubation
5. Mallampati classifications Ⅰ-Ⅱ

Exclusion Criterias:

1. Emergency operation
2. Anticipated difficult airway or history of intubation difficulties
3. Be allergic to any of the drugs used in the experiment, or have a history of drug allergy
4. Preoperative use of analgesic, sedative and other drugs
5. Uncontrolled hypertension and heart disease
6. Have a history of heavy smoking and alcohol abuse, serious drug abuse, and severe systemic infections
7. There are severe mental and nervous system symptoms, and patients cannot cooperate with the study, such as language comprehension disorder, mental illness, etc
8. Other clinical trials were conducted within 3 months prior to inclusion in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Remifentanil TCI effect site concentration | through study completion, an average of 20 min
  preestablish remifentanil TCI effect site concentration(ng/ml)

SECONDARY OUTCOMES:
mean arterial pressure | at entering the operation room(T1), at immediately before DLT intubation(T2), at immediately after DLT intubtion(T3), at 1 minute(T4)/2 minutes (T5)/3 minutes(T6) after DLT intubation
  mean arterial pressure in mmHg
heart rate | at entering the operation room(T1), at immediately before DLT intubation(T2), at immediately after DLT intubtion(T3), at 1 minute(T4)/2 minutes (T5)/3 minutes(T6) after DLT intubation
  heart rate in bpm
Narcotrend index | at entering the operation room(T1), at immediately before DLT intubation(T2), at immediately after DLT intubtion(T3), at 1 minute(T4)/2 minutes (T5)/3 minutes(T6) after DLT intubation
  Narcotrend index in Arabic numerals

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, M.D., Study Chair — alluo@tjh.tjmu.edu.cn
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No